CLINICAL TRIAL: NCT01207349
Title: Type 2 Diabetes Secondary Prevention Trial at the Reunion Island
Brief Title: Type 2 Diabetes Secondary Prevention
Acronym: RP2
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Groupe Hospitalier Sud Reunion (Other)
Responsible Party: Sponsor
Other Study IDs: RBM01-23
Record Dates: First submitted 2010-09-14; First posted 2010-09-22 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2012-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Secondary prevention; Physical activity; Nutritional education; HbA1c; Reunion island; diabetic patients, both female and male, age >=18 years, able to practise a physical activity, in Saint Pierre (GHSR) and Saint Denis (CHD)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- close follow-up by nurse: close follow-up by nurse : patients were visited each tree months
  Interventions: Behavioral: Secondary prevention intervention trial
- standard follow up: stantdard follow up at one year
  Interventions: Behavioral: standard follow up

INTERVENTIONS:
Behavioral: Secondary prevention intervention trial — Close follow-up by nurses, exercise physiologist and dieteticians
  Other Names: Rédia-prev2
  Groups: close follow-up by nurse
Behavioral: standard follow up
  Groups: standard follow up

SUMMARY:
Three hundred and ninety height diabetic patients were educated during a week of hospitalisation (nutritional and physical-activity advices). After that, they were randomized in two groups : frequent follow-up (each three month) by educational nurses and dieteticians, versus no follow-up (control group). All patients were evaluated one year after their inclusion,by HbA1c (primary outcome), anthropometry, other cardiovascular risk factors, nutritionnal and physical-activity behaviours.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes patient aged >=18 years

Exclusion Criteria:

* incapacity to a moderate physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2002-08; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
%HbA1c | at inclusion and at one year
  measure of % HbA1c at inclusion and at one year and comparison between intervention and control groups

SECONDARY OUTCOMES:
anthropometry | at inclusion and at one year
  BMI, waist, %fat mass and comparison between intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Schwager, MD, Study Director — GHSR
Locations (1):
- GHSR, Saint-Pierre, La Réunion, France

REFERENCES:
- [Result] Debussche X, Rollot O, Le Pommelet C, Fianu A, Le Moullec N, Regnier C, Boyer MC, Cogne M, Bakiri F, Schwager JC, Favier F. Quarterly individual outpatients lifestyle counseling after initial inpatients education on type 2 diabetes: the REDIA Prev-2 randomized controlled trial in Reunion Island. Diabetes Metab. 2012 Feb;38(1):46-53. doi: 10.1016/j.diabet.2011.07.002. Epub 2011 Oct 24. PMID 22030240